CLINICAL TRIAL: NCT07084701
Title: Effects of Non-Invasive Superficial Craniocervical Lymphatic Drainage (NSCLD) on Memory and Cognitive Function in Adults With Sleep Deprivation: A Proof-of-Concept Study
Acronym: NSCLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tao Liu (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor-Investigator, Tao Liu, MD, The George Institute
Organization: The George Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NSCLD
Record Dates: First submitted 2025-07-08; First posted 2025-07-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Sleep Deprivation
Keywords: Sleep Deprivation; Non-Invasive Superficial Craniocervical Lymphatic Drainage; Memory; Cognitive Function; NSCLD
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSCLD group (Experimental): NSCLD for 30 minutes, repeated after a 10-minute interval
  Interventions: Device: Non-Invasive Superficial Craniocervical Lymphatic Drainage (NSCLD)
- Control group (Sham Comparator)
  Interventions: Device: sham-intervention treatment

INTERVENTIONS:
Device: Non-Invasive Superficial Craniocervical Lymphatic Drainage (NSCLD) — Participants will be randomly assigned to either an intervention group receiving NSCLD or a control group receiving a sham-intervention treatment. Cognitive function will be assessed using standardized tests before and after the intervention.
  Arms: NSCLD group
Device: sham-intervention treatment — Participants will be randomly assigned to either an intervention group receiving NSCLD or a control group receiving a sham-intervention treatment. Cognitive function will be assessed using standardized tests before and after the intervention.
  Arms: Control group

SUMMARY:
This Effects of Non-Invasive Superficial Craniocervical Lymphatic Drainage (NSCLD) on Memory and Cognitive Function in Adults with Sleep deprivation: A Proof-of-Concept Study aims to investigate the effects of Non-Invasive Superficial Craniocervical Lymphatic Drainage (NSCLD) on memory and cognitive function in adults experiencing sleep deprivation(SD). Given the known impact of SD on cognitive performance, this study seeks to explore whether NSCLD, as a non-invasive intervention, can mitigate the cognitive impairments associated with SD.

DETAILED DESCRIPTION:
Sleep deprivation (SD) is widespread in modern society, particularly among medical students, residents, and individuals in high-stress occupations. Numerous studies have demonstrated that acute sleep deprivation significantly impairs cognitive processes such as attention, working memory, and executive function. Even short-term cognitive impairment can have serious consequences, including impaired judgment, slowed reaction times, and increased error rates.

Currently, interventions targeting cognitive decline following sleep deprivation are limited. Common strategies primarily include medications (such as caffeine and modafinil) and restorative sleep. However, these methods have limitations in both clinical and real-life settings: on one hand, medications may lead to tolerance and side effects, and on the other hand, restorative sleep often cannot reverse cognitive impairment in the short term. Therefore, developing a safe, convenient, and rapidly effective non-pharmacological intervention is of great significance.

In recent years, the glymphatic system has garnered increasing attention. This system is believed to play a key role in clearing metabolic waste from the brain, regulating sleep structure, and maintaining neurocognitive function. Superficial craniocervical lymphatic drainage (SCLD) has been proposed as a potential mechanism to improve cognitive function by enhancing the flow of cerebrospinal fluid (CSF) and lymph, reducing neuroinflammation, and minimizing the accumulation of metabolic waste.

In June 2025, a study published in Nature provided the first in vivo evidence supporting this hypothesis. Researchers applied non-invasive mechanical stimulation to the superficial lymphatic system on the skin surface of the mouse neck, resulting in a doubling of CSF drainage efficiency to cervical lymph nodes and correction of impaired brain-lymphatic efflux function in aged mice. These findings provide direct mechanistic support for the potential application of non-invasive SCLD intervention in humans.

Therefore, this study aims to establish an acute sleep deprivation model in healthy adults and explore the immediate effects of NSCLD intervention on cognitive function, with the goal of providing preliminary clinical evidence for non-pharmacological intervention strategies related to the brain-lymphatic pathway.

ELIGIBILITY:
Inclusion Criteria:

* College student ≥18 years, all of whom have passed a standardized entrance examination;
* No failed exams during the course of study;
* Sleep deprivation;
* In good health, with no mental or psychological disorders;
* No recent use of medications that may affect memory and cognition;
* Voluntary participation and able to undergo cognitive function and memory testing;
* Informed consent provided

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Presence of acute or chronic medical conditions (e.g., severe hypertension, diabetes, cardiovascular disease) that could confound the results.
* History of craniocervical trauma or surgery.
* Current use of sedative or anxiolytic medications that could influence sleep or cognitive function.
* Participants who are unable to follow the procedures or complete the assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Digit Span Test | Day 1 (Baseline) and Day 2, repeat after a 2-week washout period
  Evaluate memory function. 1 point for each correct string of numbers. Total score: forward score + backward score. Higher scores mean a better outcome.
Montreal Cognitive Assessment (MoCA) | Day 1 (Baseline) and Day 2, repeat after a 2-week washout period
  The maximum score is 30 points. ≥26 points is normal. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Changes in anxiety, stress, irritability, etc. before and after instant massage | Day 1 (Baseline) and Day 2, repeat after a 2-week washout period
  use Multidimensional VAS Battery. 0 points are "not at all", and 100 points are "extremely strong" (points 0- 100)
Brain metabolic markers and other metabolic indicators | Day 1 (Baseline) and Day 2, repeat after a 2-week washout period
  Collect blood for analysis of Aβ42/40, T-Tau, p-tau217, Plasma cortisol, Salivary α-Amylase and β-Endorphin.
EEG power in alpha, beta, delta and theta band | Day 1 (Baseline) and Day 2, repeat after a 2-week washout period
  Measure the power of different frequency bands of EEG and compare the changes.
Heart rate variability (HRV) | Day 1 (Baseline) and Day 2, repeat after a 2-week washout period
  Analyze the different indicators of HRV, including RMSSD, LF, HF, LF/HF ratio, SDNN, etc.
modified TOEFL iBT | Day 1 (Baseline) and Day 2, repeat after a 2-week washout period
  Developed by English language professionals based on TOEFL difficulty and standards, with self-compiled test papers. Full marks: 100 points. To evaluate working memory, learning memory, attention allocation, information processing speed, executive functions (such as planning and monitoring), and the retrieval and integration of long-term memory, among other aspects.
Computerized Cognitive Assessment | Day 1 (Baseline) and Day 2, repeat after a 2-week washout period
  Use N-back task and Psychomotor vigilance task (PVT) ,measure metrics such as reaction time and accuracy rate.
Functional magnetic resonance imaging (fMRI) | Day 1 (Baseline) and Day 2, repeat after a 2-week washout period
  Using functional magnetic resonance imaging to evaluate brain functional activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided